| IRB Approval Date |
|-------------------|

**Title of research study:** Medical Marijuana Use and Driving Performance: A Test of Psychomotor Function in Adults 50 and Older

Investigator: Nicole Ennis, PhD

**<u>Key Information</u>**: The following is a short summary of this study to help you decide whether or not to be a part of this study. More detailed information is listed later on in this form.

#### Why am I being invited to take part in a research study?

We invite you to take part in a research study because you are starting medical marijuana. Your participation will help us examine the risks and benefits of medical marijuana as it relates to psychomotor function and driving ability.

### What should I know about a research study?

- Someone will explain this research study to you.
- Whether or not you take part is up to you.
- You can choose not to take part.
- You can agree to take part and later change your mind.
- Your decision will not be held against you.
- You can ask all the questions you want before you decide.

### Why is this research being done?

The purpose of this research study is to examine the relationship between medical marijuana use and psychomotor function in adults 50 and older.

## How long will the research last and what will I need to do?

We expect that you will be in this research study for 3 months and 1 week. The entire participation time will require about 3 hours to complete over the course of 3 months and 1 week. This will consist of 3 sixty-minute meetings with study team members over the course of 3 months and 1 week.

More detailed information about the study procedures can be found under "What happens if I say yes, I want to be in this research?"

# Is there any way being in this study could be bad for me?

There may be questions that you may find unpleasant or difficult to answer. Questions will include things such as drug use, pain, and depression. You may refuse to answer any question. We will try to answer any questions you have and discuss any concerns you may have about answering a question. If you are unsure of any of the questions, you may ask the interviewer to explain them. More detailed information about the risks of this study can be found under "Is there any way being in this study could be bad for me? (Detailed Risks)"

Will being in this study help me in any way?

There are no direct benefits to you for taking part in this research study.

### What happens if I do not want to be in this research?

Participation in research is completely voluntary. You can decide to participate or not to participate.

Your alternative to participating in this research study is to not participate.

### What are the informed consent requirements related to ClinicalTrials.gov?

A description of this clinical trial will be available on <a href="http://www.ClinicalTrials.gov">http://www.ClinicalTrials.gov</a>, as required by U.S. Law. This Web site will not include information that can identify you. At most, the Web site will include a summary of the results. You can search this Web site at any time.

**<u>Detailed Information:</u>** The following is more detailed information about this study in addition to the information listed above.

#### Who can I talk to?

If you have questions, concerns, or complaints, or think the research has hurt you, talk to the research team at Nicole Ennis, PhD, Principal Investigator, 850-644-7955.

This research has been reviewed and approved by an Institutional Review Board ("IRB"). You may talk to them at 850-644-7900 or humansubjects@fsu.edu if:

- Your questions, concerns, or complaints are not being answered by the research team.
- You cannot reach the research team.
- You want to talk to someone besides the research team.
- You have questions about your rights as a research subject.
- You want to get information or provide input about this research.

## How many people will be studied?

We expect about 60 people total will be in this research study.

# What happens if I say "yes" to being in this research?

First, you will be asked to participate in a battery of tests, including psychosocial measures and a cognitive test. Next, you will be asked to provide a urine specimen that will be used to detect the presence or absence of THC and other drugs. Finally, you will be asked to participate in an approximately 5-minute simulator adaptation drive and an approximately 10-minute main drive. We will monitor you for symptoms of simulator sickness before, during, and after the drives. Additionally, we will also request permission to extract needed data on an ongoing basis from your electronic medical records for a period of 12 months after your enrollment in the study.

Mandatory Reporting: Florida law requires that all study staff must report any reports of child abuse, suicidal or homicidal behaviors to the appropriate authorities. These include physical injury to any child not caused by an accident or information that tells staff a person is in danger of physical harm. If you report that you may harm yourself or others you may be referred for immediate care. If you have any questions now or at any time during the study, please contact one of the research team members listed in question 3 of this form.

# What are my responsibilities if I take part in this research?

We will contact everyone by phone and ask you to meet with us again both 1 and 3 months after your first meeting with the study team member for an in-person meeting. During these meetings we will ask you to repeat the simulated drive from the first session, including an approximately 5-minute simulator adaptation drive and an approximately 10-minute main drive. We will also administer the same questionnaire from the first session and collect another urine sample.

Also, please be aware that driving a real-life, non-simulated vehicle while under the influence of marijuana is driving under the influence (DUI) in Florida, and is illegal. Therefore, if you decide to participate in this research, you are solely responsible for ensuring that you are not under the influence of any substances or experiencing any drug-related effects when driving to or from the University

campus for your study visits. It may be necessary to arrange for someone else to drive you to these visits or use public transportation, taxi or ride-sharing services.

# What happens if I say "yes," but I change my mind later?

You can leave the research at any time it will not be held against you.

If you stop being in the research, already collected data may not be removed from the study database. You will be asked whether the investigator can collect data from your routine medical care. If you agree, this data will be handled the same as research data.

# Is there any way being in this study could be bad for me? (Detailed Risks)

- Psychological risks. Participants may find some questions difficult to answer and it may embarrass them or make them uncomfortable. We have trained the people gathering data to explain why the question is being asked if needed and you can refuse to answer any question.
- Privacy risks and Legal Risks. There is the potential that privacy could be breached. However, this is not likely as all data and computer files will be stored in a locked, secure area, and will only be accessed by authorized personnel. Photocopies of original records and computer files will be deidentified and labeled with a unique subject identifier. Therefore, all assessment instruments and related study data will be identified by number only. All research questionnaires will be stored in locked file drawers or on a secure server accessible only to research staff. To provide additional data security a master key linking identifying participant information with the study number will be secured in a different locked file.
- Economic risks. If privacy is breached it could impact your ability to obtain employment. However, this is not likely as all data and computer files will be stored in a locked, secure area, and will only be accessed by authorized personnel.

You and your insurance company will be charged for the health care services that you would ordinarily be responsible to pay. In some cases, insurance will not pay for services ordinarily covered because these services were performed in a research study. You should check with your insurance to see what services will be covered by your insurance and what you will be responsible to pay.

# What happens to the information collected for the research?

Efforts will be made to limit the use and disclosure of your personal information, including research study and medical records, to people who have a need to review this information. We cannot promise complete secrecy. Organizations that may inspect and copy your information include the IRB and other representatives of this organization and the National Institute on Drug Abuse.

Mandatory Reporting: Florida law requires that all study staff must report any reports of child abuse, suicidal or homicidal behaviors to the appropriate authorities. These include physical injury to any child not caused by an accident or information that tells staff a person is in danger of physical harm. If you report that you may harm yourself or others you may be referred for immediate care. If you have any questions now or at any time during the study, please contact one of the research team members listed in question 3 of this form.

If identifiers are removed from your identifiable private information or identifiable samples that are collected during this research, that information or those samples could be used for future research studies or distributed to another investigator for future research studies without your additional informed consent.

The sponsor, monitors, auditors, and the IRB will be granted direct access to your medical records to conduct and oversee the research. By signing this document, you are authorizing this access.

We may publish the results of this research. However, we will keep your name and other identifying information confidential to the extent allowed by law.

## Can I be removed from the research without my OK?

The person in charge of the research study or the sponsor can remove you from the research study without your approval. Possible reasons for removal include participant is a danger to self or others, has lost cognitive capacity to participate.

#### What else do I need to know?

This research is being funded by the National Institute on Drug Abuse

If you agree to take part in this research study, we will pay you \$50 for each assessment, which is a total of \$150 if all 3 assessments are complete for your time and effort.

MOD00001150 FSU IRB Approved 9 April 2021

# Permission to Take Part in a Human Research Study

# **Signature Block for Capable Adult**

Your signature documents your permission to take part in this research.

Signature of subject

Printed name of subject

Signature of person obtaining consent

Printed name of person obtaining consent

IRB Approval Date